CLINICAL TRIAL: NCT03864016
Title: Ability of Pupillometry to Reduce Sufentanil Consumption in Planned Cardiac Surgery: Randomized, Controlled, Single-center Clinical Superiority Trial
Acronym: PUCCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BERTHOUD 2018
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Patients Undergoing Cardiac Surgery; Patients With Coronary Artery Bypass Surgery With CEC
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Other)
  Interventions: Drug: Induction and maintenance of anesthesia; Drug: Adaptation of sufentanil doses according to the usual protocol
- Pupillometry group (Experimental)
  Interventions: Drug: Induction and maintenance of anesthesia; Drug: Adjustment of sufentanil doses according to pupillometry

INTERVENTIONS:
Drug: Induction and maintenance of anesthesia — The hypnotic agent used is Propofol and the morphine agent used is Sufentanil.
Drug: Adaptation of sufentanil doses according to the usual protocol — At induction the target concentration of sufentanil is 0.5 ng/ml. The sufentanil dose is decided by the anaesthetist, taking into account the operating times (induction, TIO, incision, opening and sternal spacing, CEC, closure), the usual data provided by the monitoring: heart rate, blood pressure, BIS, EtCO2, modification of insufflation pressures.
  Arms: Standard group
Drug: Adjustment of sufentanil doses according to pupillometry — At induction, the target concentration of sufentanil is 0.5 ng/ml. The dose of sufentanil is then adjusted according to the dilation reflex obtained with the PPI (Pain Pupillary Index) at predefined times.
  Arms: Pupillometry group

SUMMARY:
The objective of general anesthesia is to obtain a loss of consciousness, stillness, and sufficient analgesia to allow surgery. Thus, general anesthesia has two components: hypnosis and analgesia. Combining these two components, with parallel use of a hypnotic agent and a morphine agent makes major surgery possible by limiting the stress on the body. In clinical practice, hypnosis can be assessed by a monitor of the depth of BIS®-type anesthesia, based on a simplified measurement of the patient's spontaneous cortical electroencephalographic activity. However, BIS® type monitors do not specifically judge analgesia.

Traditionally, analgesia is assessed on the basis of hemodynamic changes (blood pressure, heart rate) in relation to a nociceptive stimulus. There is an interaction between pain and cardiovascular control that is mediated by the baroreflex system. But not all hemodynamic changes during general anesthesia are necessarily secondary to nociceptive stimulation. For example, hypovolemia may be responsible for tachycardia without causing pain; opening the pericardium during cardiac surgery may increase blood pressure by increasing cardiac output.... On the other hand, a decrease in hemodynamic response can be observed in relation to the depressant effect of anesthetic agents, despite a lack of analgesia. Similarly, patients' disease-modifying treatments may mask hemodynamic responses (e.g. beta blocker). Thus, the appearance of tachycardia or high blood pressure during surgery does not necessarily reflect a nociceptive process. Currently, the available data do not allow the anaesthetist to differentiate between real hemodynamic changes related to nociception and sympathicotonia. This leads to typical management consisting of an increase in the dosage of morphine.

Pupillometry (monitoring the pupillary dilation reflex) is a simple and sensitive clinical approach that can be done during general anesthesia to specifically monitor the nociceptive component. The main objective of monitoring is to achieve a more rational use of opioids. This means optimizing opioid dosing, ensuring safety by monitoring the lowering of opioid dosages intraoperatively without the risk of waking up, and reducing postoperative hyperalgesia. In the context of cardiac surgery, the interpretation of hemodynamic changes could be facilitated by nociception monitoring coupled with anesthesia monitoring (BIS). Reducing opiod doses without changing other clinical parameters could ensure better hemodynamic stability in increasingly fragile patients.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given written consent
* Adult patient
* Patient undergoing coronary artery bypass surgery with CEC, with or without valve surgery, by sternotomy.
* ASA <4.

Exclusion Criteria:

* Person not affiliated to the national health insurance system
* Person subject to legal protection (curatorship, guardianship)
* Person who has been deemed mentally incompetent
* Pregnant, parturient or breastfeeding woman
* Adult unable or unwilling to provide consent
* Patient with preoperative cognitive dysfunction (MMS <13) (APPENDIX 6),
* Patient with morphine intolerance,
* Patient on long-term opioid treatment,
* Emergency surgery,
* Eye disease, corneal injury, or wearing contact lenses, a neurological disease that can influence the pupillary reflex,
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Total dose of sufentanil required per operation | Through study completion an average of 2 years
  Total dose of sufentanil expressed in µg

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Berthoud V, Nguyen M, Appriou A, Ellouze O, Radhouani M, Constandache T, Grosjean S, Durand B, Gounot I, Bahr PA, Martin A, Nowobilski N, Bouhemad B, Guinot PG. Pupillometry pain index decreases intraoperative sufentanyl administration in cardiac surgery: a prospective randomized study. Sci Rep. 2020 Dec 3;10(1):21056. doi: 10.1038/s41598-020-78221-5. PMID 33273644